CLINICAL TRIAL: NCT00317525
Title: Effects of Different Add Powers on the Comfort and Productivity of Computer Users With Fixed or Free Head Movement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Optometric Association (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: X050314015
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2005-05

CONDITIONS: Refractive Errors; Asthenopia
Keywords: Refractive error; Asthenopia
MeSH Terms: conditions — Refractive Errors; Asthenopia

INTERVENTIONS:
Device: Spectacle Lenses

SUMMARY:
The aim of this study is to examine the relationship between optical blur from poor refractive corrections (glasses) of older workers using computers and their productivity and comfort in the workplace. The investigators believe that improving the visual status of subjects who use computers will have a beneficial effect on productivity and visual comfort.

DETAILED DESCRIPTION:
The aim of this study is to examine the relationship between optical blur from poor refractive corrections (glasses) of older workers using computers and their productivity and comfort in the workplace. We believe that improving the visual status of subjects who use computers will have a beneficial effect on productivity and visual comfort. All subjects will be required to complete a vision screening at no charge to decide if they qualify for the study. This is a double-blind study, which means that neither the subject nor the doctors will know which pair of lenses you will be wearing during the parts of the study. Subjects will complete a total of 4 hours of testing. The total amount of testing will be divided into ten 15-minute periods. During each period, the investigator will place different lenses in a trial frame. The trial frame that the subject will wear during the experiment will have their prescription for near plus an unknown pair of lenses. During the testing, the subject will complete a task involving finding and deleting apostrophes from a manuscript on a standard computer. Either the investigator or co-investigator will explain how to do this simple task. Subjects will answer a short survey before and after these tasks to check on symptoms resulting from using the computer. The following periodic measurements will be made during the study: productivity and accuracy to search for apostrophes (') in a document on one of the states of the U.S. These tasks will require a total of 4 hours testing with a total of ten pairs of trial lenses during a single visit.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or greater
* 20/40 visual acuity or better in each eye
* Use a computer at least 1 hour per work day

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2005-05; Study Completion 2006-06

PRIMARY OUTCOMES:
Visual comfort
Productivity (correct words per hour)

CONTACTS AND LOCATIONS:
Overall Officials: Kent M Daum, O.D., Ph.D., Principal Investigator — School of Optometry, University of Alabama at Birmingham
Locations (1):
- School of Optometry, Birmingham, Alabama, United States